CLINICAL TRIAL: NCT05271864
Title: Accuracy of Apple Watch to Measure Cardiovascular Indices in Patients With Chronic Diseases: A Cross Sectional Study
Brief Title: Smart Watch, Heart Rate and So2 in Chronic Patients
Status: Completed | Type: Observational
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Alaa Khushhal, Principal Investigator, Umm Al-Qura University
Other Study IDs: HAPO-02-K-012-2022-02-959
Record Dates: First submitted 2022-02-17; First posted 2022-03-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Chronic Disease
Keywords: Oxygen saturation; Heart rate; diabetes mellites; Hypertension; hyperlipidemia
MeSH Terms: conditions — Chronic Disease; Hypertension; Hyperlipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: diabetes mellites
  Interventions: Device: Apple Watch
- Group B: hypertension
  Interventions: Device: Apple Watch
- Group C: hyperlipidemia
  Interventions: Device: Apple Watch

INTERVENTIONS:
Device: Apple Watch — Apple Watch

SUMMARY:
Background: Apple watch validity to measure the heart rate (HR) and oxygen saturation (Spo2) in healthy subjects has been investigated, but its accuracy and validity for patients with chronic non-communicable diseases such as diabetes mellites (DM), hyperlipidemia and hypertension (HTN) is still unclear. Patients with chronic diseases as DM, HTN and hyperlipidemia who have hypoxemia are advised to continuously monitor their Spo2. Therefore, this study aims to investigate the accuracy of the Apple watch in measuring the Spo2 and heart rate in patients with chronic diseases.

Method: A cross sectional study will invite ninety-five patients with chronic diseases to participate in this study and the eligible participants will be allocated into three groups. The first group (Group-A) will include patients with the DM, the second group (Group-B) will include the patients with HTN and the third group will include patients with hyperlipidemia. All participants will use the apple watch to evaluate the Spo2 against the pulse oximeter at rest. The main outcome will be the Spo2 and heart rate that will be evaluated at rest and before and after exercise for 15 minutes using the Apple watch, Spo2 and Polar HR monitored using the pulse oximeter.

DETAILED DESCRIPTION:
Introduction:

Assessment of the heart rate (HR) is an essential process to determine proper exercise training intensity. (1) Utilization of the 12-leads electrocardiogram (ECG) is considered most objective heart rate assessment procedure. Polar chest strap arises as an alternative to the ECG when it is not accessible to use it outside the laboratories. The Polar chest strap proved valid and reliable instrument when tested against the ECG in healthy subjects (2-4) and patients with cardiac diseases (5) at rest and during training. Monitoring the resting as well as the post-training heart rate (heart rate recovery) is essential because it helps predicting the cardiopulmonary fitness level as well as the mortality risk among evaluated personnel. (6)

Diabetes mellitus is a rapidly growing non-communicable chronic disease worldwide, becoming one of the most alarming health problems in the 21st century. The overall estimated prevalence of diagnosed diabetes in 2018 was 26.9 million US subject of all ages (8.2% of the US population) (7) The International Diabetes Federation (IDF) has estimated the total number of persons with DM across the world will rise from 536.6 million in 2021 to 783.2 million by 2045, with about 94% of the increase in the number of subjects with diabetes by 2045 will be within the low and middle-income countries. The global incidence also projected to increase from 16.3% in 2021 to 19.2% by 2025 in middle- and low-income countries. The prevalence of diabetes in adults (20-79 years old) in the Middle East and North Africa was estimated to be 16.2% compared to 19.3% in 2045. (8) Hypertension possess significantly increased public health risk and population challenge. The prevalence of hypertension was 6.0, 4.2 and 4.9% in male, female and all subjects, respectively. (9) Hypertension prevalence is increasing in KSA, the rate exceeds 25% among the adult Saudi subjects. Monitoring the hypertension-related disturbances is an urgent concept to prevent its organs-damaging. (10) Regional study at Majmaah, Saudi Arabia reported that the hypercholesterolemia prevalence was 45.3%, with no significant difference between both genders. (11) A study by Al-Nozha et al., reported that the hyperlipidemia continues reaching higher prevalence rate recently. The hypercholesterolemia prevalence among the 30-70 years old subjects reached 54.9% and 53.2% for males and females respectively, Hypertriglycemia prevalence was 47.6% in male compared to 33.7% in females. (12) More recently; a study by reported that the prevalence of Hypercholesterolemia among Saudi population ≥ years old is around 12.5%, with males have higher rate (56.7%) compared to females who have lower s rate (43.3%). Close monitoring of the vital signs and cardiovascular variables in patients with chronic non-communicable diseases is indicated since many harmful consequences can be prevented via increasing community awareness and education. (13) Diabetes Mellitus is chronic debilitating disorder requires well-organized efforts and continuous monitoring to limit the impact of disease-associated hazards and long-term complications. (14) The process of SpO2 evaluation is important because it indirectly reflects the subject's organs oxygen requirements. The traditional SpO2 measuring procedure is invasive and painful, requiring collection and assay of arterial blood sample using a blood gas analyzer. (15) Previous trials proposed evaluating the SpO2 non-invasively using simple procedure, with keeping maximum accuracy. (16) Pulse oximetry is a well-known noninvasive instrument used for monitoring and evaluation of SpO2). (17) Routine and frequent screening of patients with chronic diseases is recommended especially with age over 50 years and presence of other comorbidities as HTN and hyperlipidemia. (18) Pulse oximetry is used to measure the level of the SpO2, with low blood flow is associated with lower SpO2. (19) The HR is tightly and linearly correlated with the oxygen consumption at specified time point.(20) Monitoring of other vital variables as the oxygen saturation (SpO2) is recommended in patients suffering hypoxia to improve their survival, (21) as in post-operative and post-arrest cardiac patients, (22) with the pulse oximeter is the widely used instrument to evaluate the SpO2 because of accuracy and ease of application. (23) Quiet recently; the Apple smart watch appeared as a new tool to measure the HR. all the Apple watch versions can monitor the HR, but the blood SpO2 can be only measured by only the latest 6 and 7 versions. The concept of utilizing the Apple watch to measure the HR depends on the Photoplethysmography (PPT) non-invasive measurement procedure applied using wrist-worn watch that continuously monitors both heart beats and blood color changes over time. The PPT is a commonly used approach to measure the cardiac output, blood pressure and SpO2 in verities of medical instruments, (24) that can help discovering the cardiovascular insults and complications at early stages. (25) Implemented new technology and updated features that enable the Apple watch to monitor the HR is available only in updated series-6 and 7. Very limited number of studies evaluated the validity of the Apple watch against pulse oximeter in measuring the SpO2 (the Spo2 was evaluated in 23 patients with chronic obstructive pulmonary disease, 61 patients with interstitial lung diseases and 16 health control subjects). the Apple watch results showed strong positive correlations with that of the pulse oximeter (r=0.81, P<0.0001), furthermore; this study recommended testing the Apple watch validity for measuring the SpO2 in other groups of patients. (26) The Apple watch is a smart instrument with advanced technology measuring the Spo2 and heart rate but its validity in patients with chronic diseases including patients with diabetic mellites, hypertension and hyperlipidemia is still unknown. Therefore, this will be the first study to evaluate the Apple watch accuracy and validity in measuring the Spo2 and heart rate in patients with chronic diseases including diabetic mellitus, hypertension, hyperlipidemia.

Method:

A cross sectional study will be conducted, ninety-five chronic patients will be invited to participate in this study. The study design will be in form of 3-groups: first group will include 35 patients with diabetes and the second group will include 35 patients with hypertension. The third group will be around 35 patients with hyperlipidemia. The distribution of patients and number of groups will be based on the availability of the patients with chronic non-communicable diseases at Umm Al-Qura University Medical Center. All participants in this study will wear the Polar chest strap HR and the Apple Watch at rest, during short session of mild to moderate intensity exercise [50-70% (maximum heart rate-Resting heart rate) + resting heart rate] for 15 minutes and after exercise. The pulse oximeter will be used at rest (pre) and after exercise.

Under resting condition; the pulse oximeter will be fitted on a warm finger while the participant assumes setting position, with the patient in the upright (sitting) position and resting. The SpO2 reading will be recorded after being stabilized on the pulse oximeter instrument. (27, 28) The exercise session will be about 15-minutes duration at mild to moderate intensity according to the heart rate reserve (HRR) using the treadmill and the cycle ergometer, preceded by a 3-minutes warm-up, and followed by 3-minutes cool-down. The HR will be recorded every 30 seconds during whole period and the oxygen saturation will be recorded five times at rest and after exercises.

This study will follow the Declaration of Helsinki 1975 principles, revised in 2000 and will be conducted at the Umm Al-Qura University Medical Center, and will be in line with the Faculty of Applied Medical Sciences, Umm Al-Qura University ethical guidelines. Each participant will sign a written consent approving the volunteer participation in this study and agreeing for publication of its results. Suitable sample size was be computed using the online G-power tool (https://download.cnet.com/G-Power/3000-2054_4-10647044.html), considering the effect size = 0.5, giving a sample size of 54 participants to provide reliable results. Extra-number will be included to substitute any participant's withdrawal or discontinuation.

Inclusion criteria: eligible participants will be patients with chronic diseases as those with stable diabetes mellitus type 1 or 2, hypertension but not more than 180 mm.Hg and patients with hyperlipidemia.

Exclusion criteria: patients with uncontrolled diabetes mellitus, uncontrolled hypertension and hyperlipidemia will be all excluded from the study. Also, patient with other disease rather than that described in the inclusion criteria will be also excluded.

Risk management:

All measurements in this study will be done as the normal measurements for each patient with chronic non-communicable disease who visited the Umm Al-Qura University Medical Center, so there is no risk for the patients to take part in this study. In case any terribly ill happen because of the study procedure, the cardiologist (Dr. Mahmoud) will supervise each patient in this study.

Data analysis:

All data will enter into the SPSS program for analyses. First, a descriptive analysis will be performed to show results in form of means and standard deviations. The results of this study will be analyzed using the Pearson correlation test to test the difference between the apple watch and the Pulse oximeter in measuring SpO2 and heart rate in measuring heart rate to test Apple watch validity. The P value will be set at 0.05 for significant results.

ELIGIBILITY:
Inclusion Criteria:

* eligible participants will be patients with chronic diseases as those with:
* Stable diabetes mellitus type 1 or 2.
* Hypertension but not more than 180 mm.Hg
* Hyperlipidemia

Exclusion Criteria:

* patients with :
* Uncontrolled diabetes mellitus.
* Uncontrolled hypertension.
* Uncontrolled hyperlipidemia will be all excluded from the study.
* Patient with other chronic diseases rather than that described in the inclusion criteria will be also excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic mellites, hypertension and hyperlipidemia
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation | over 10 minutes at rest
Oxygen Saturation | over 10 minutes after exercise

SECONDARY OUTCOMES:
Heart rate | over 31 minutes
  Heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Umm Al-Qura medical center, Al Makhwāh, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
May be for publication in the article

REFERENCES:
- [Derived] Khushhal AA, Mohamed AA, Elsayed ME. Accuracy of Apple Watch to Measure Cardiovascular Indices in Patients with Chronic Diseases: A Cross Sectional Study. J Multidiscip Healthc. 2024 Mar 11;17:1053-1063. doi: 10.2147/JMDH.S449071. eCollection 2024. PMID 38496326